CLINICAL TRIAL: NCT03877991
Title: Bioequivalence Assessment of Cannabidiol (CBD) Administrated in Oral Formulations
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0352-18-HMO-CTIL
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: Bioavailability; Pharmacokinetics
MeSH Terms: conditions — Pain | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Randomized Open Label, three way cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD-sesame oil capsule (Experimental): 12 volunteers will receive a single oral dose of CBD in a sesame oil vehicle filled in a capsule, with 200 mL of water. The dose of CBD to be administrated is 90 mg.
  Interventions: Drug: CBD-sesame oil capsule
- CBD-LNL capsule (Experimental): 12 volunteers will receive a single oral dose of CBD-LNL formulation filled in a capsule, with 200 mL of water. The dose of CBD to be administrated is 90 mg.
  Interventions: Drug: CBD-LNL capsule
- CBD powder form capsule (Experimental): 12 volunteers will receive a single oral dose of CBD in powder form filled in a hard gelatin capsule, with 200 mL of water. The dose of CBD to be administrated is 90 mg.
  Interventions: Drug: CBD powder form capsule

INTERVENTIONS:
Drug: CBD-sesame oil capsule — A capsule containing cannabidiol dissolved in sesame oil and surfactant vehicle.
  Other Names: Cannabidiol in sesame oil vehicle cpausle
  Arms: CBD-sesame oil capsule
Drug: CBD-LNL capsule — A capsule containing Cannabidiol dissolved in self nano emulsifying formulation
  Other Names: Cannabidiol in Long Chain Nano Lipospheres formulation
  Arms: CBD-LNL capsule
Drug: CBD powder form capsule — Powder of Cannabidiol filled in a hard gelatin capsule, without formulation.
  Other Names: Cannabidiol solid dosage form
  Arms: CBD powder form capsule

SUMMARY:
The oral bio-availability of cannabidiol (CBD) is low due to poor water solubility and susceptibility to extensive first pass metabolism, resulting in relative bio-availability of 6%.This project is designed to evaluate the plasma concentration vs. time profile of a self emulsifying drug delivery system termed Long Chain Nano Lipospheres (LNL) for enhancing the oral bio-availability of cannabidiol (CBD). The main goal of this study is to evaluate the bio-equivalence of CBD in the LNL product, compared to CBD in a sesame oil vehicle and CBD without any formulation, in powder form. Bio-equivalence is measured by AUC 0-24h, Tmax and Cmax.

DETAILED DESCRIPTION:
Cannabidiol (CBD) is considered the non-psychoactive component of the cannabis plant with a myriad of pharmacological attributes. There is preliminary data that CBD can be a useful treatment for different therapeutic conditions such as epilepsy, anxiety, pain etc. CBD has been investigated for its analgesic effect in patients with neuropathic and chronic pain, especially resistant to other treatments. Further supportive evidence for CBD's efficacy in treatment of pain, is established pre-clinically and requires additional research in a clinical setting. The use of CBD in epilepsy has been assimilated in treatment guidelines in many countries including Israel. However, the potential medical use of whole-plant cannabis extracts, particularly in children with a developing brain, is limited by the psychoactive properties and the adverse effects associated with long-term THC use.

Although a therapeutic rational for the use of CBD has been demonstrated, an optimal oral dosage form to deliver this compound is not available yet. Oral administration is challenging because of CBD's poor solubility and extensive first pass metabolism, leading to an oral bioavailability of approximately 6%.

In this project, investigators utilize a bio-pharmaceutical method to enhance the bioavailability of CBD using an advanced self-emulsifying drug delivery system termed Long Chain Nano Lipospheres (LNL). The LNL formulation is composed of long chain triglycerides, surfactants and co-solvent. This constellation is termed the pre-concentrate, which dissolves CBD in its lipid core and administered in a soft gelatin capsule. When reaching the aqueous phase of the GI tract, this pre-concentrate spontaneously forms a drug encapsulated O/W nano emulsion. Previously, investigators have shown in a pre-clinical investigation that incorporation of CBD into the LNL is a promising strategy to increase the compound's bioavailability.

The primary goal of this study is to evaluate the bioequivalence of the developed CBD-LNL product to CBD in a sesame oil vehicle and CBD in powder form. Sesame oil is the commonly used vehicle for cannabinoids oral uptake for lack of other options. However, this option often leads to significant inter and intra subject variability in cannabinoids' plasma concentrations.

The study will be performed on 12 healthy male volunteers. It will be randomized, open label three way cross-over study intended to evaluate the pharmacokinetics of CBD. Each volunteer will receive CBD-LNL capsule, CBD in sesame oil vehicle capsule and CBD without any vehicle in powder form. All study groups will receive the same dose of CBD-90 mg. Blood samples will be drawn from forearm 30 minutes before (pre-dose) and every 30 minutes interval for the first 4 hours, then samples will be taken at 5,6,7,8,12 and 24 hours after the intake of the study drug. Blood concentration profiles of CBD and its main metabolites 7-hydroxy-CBD and CBD-glucoronide-11 will be determined in order to calculate the pharmacokinetic parameters of CBD.

The secondary study objectives is to examine pharmacodynamic (PD) variables of the developed CBD-LNL product to CBD in a sesame oil vehicle and CBD in powder form.

In order to assess the pharmacodynamic variables all study participants will be requested to undergo an experimental pain test: cold pressor test.

Cold pressor test model: During each pain cycle, the non-dominant hand is immersed in ice cold water up to the elbow over 2 minutes. Using the dominant hand, the computerized VAS device is manipulated by the subject to record the on-line VAS pain score at intervals of approximately 10 seconds. The area under the curve of the VAS pain score against time curve is determined electronically. If the hand has to be removed due to intolerable pain, this is taken as a VAS of 100 at that time point.

The test will be conducted upon arrival and at 0.5h, 1h, 2h, 3h, 4h , 6h, 8h after arrival at the clinic and completed at study cycles 1,2,3.

Study participants will also be requested to fill out a computerized test called "Alertness". The subject will be asked to press a button whenever an X appears on the screen. Which will be completed on all study cycles 1,2,3. This assessment will be performed at the following times, upon arrival at clinic, 0.5 h, 1h , 2h, 3h, 4h, 6h and 8h after arrival at clinic.

Furthermore, an additional control group- follow-up visit, will be added to this trial, in order to assess study participants pharmacodynamic (PD) variables, when subjects are not under any stress.

Control group will consist of all study subjects who will be asked to come for an additional follow -up visit during which their pharmacodynamic (PD) variables will be assessed.

During this follow up visit study participants will be requested to undergo an experimental pain model test-cold pressor test (CPT) upon arrival and at 0.5h, 1h, 2h, 3h, 4h , 6h, 8h after arrival at the clinic, as completed at study cycles 1,2,3.

Study participants will be requested to fill out a computerized test called "Alertness". The subject will be asked to press a button whenever an X appears on the screen as completed on previous study cycles 1,2,3. This assessment will be performed at the following times, upon arrival at clinic, 0.5 h, 1h , 2h, 3h, 4h, 6h and 8h after arrival at clinic.

Vital signs monitoring will also be measured for all study participants at this follow-up visit upon arrival at clinic and at 30 min, 1 h, 2 h, 3h, 4h, 6h, 8h following arrival. These measurements will be compared to participants hemodynamic measurements assessed from cycle 1,2, and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 through 45 years of age with body mass index in the range of: 19 through 30 kg/m2.

2. Participants should be able to ingest and absorb oral medications.

3. Subjects must be in good health as determined by medical history, vital signs measurements, physical examination (routine examination performed by the general physician), and clinical laboratory tests (blood count and biochemistry conducted in the Health maintenance organization in Israel( "kupat holim").

4. Potential participants will undergo a screening/explanatory interview in which their compatibility will be examined. The screening interview will be held prior to the first day of trial (at least during the near month preceding the first day of trial).

5. Subjects must be able to understand and comply with the requirements of the study (e.g. all medication, dietary, and alcohol restrictions).

6. Subjects must provide written informed consent to participate in the study after reading the information and consent form, and after having an opportunity to discuss the study with the investigator.

7. Subjects must complete the screening process within 4 weeks prior to the admission visit.

Exclusion Criteria:

1. Previous participation in an research trial involving administration of any of the investigated compounds within one month prior to the current study.
2. The subject is suffering from, or has a clinically significant history of, one or more of the following: impaired glucose tolerance, diabetes mellitus, renal disease, edema, stroke or neurological disorder, rheumatological disorder (including arthritis, joint or tendon abnormalities), pulmonary disorder (including a personal history of asthma, but excluding resolved pediatric asthma), hepatic disorder, has a personal history of seizures, history of psychosis any addictive or other psychiatric disease disorder or a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject by participation in the study.
3. The subject has a known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) 1 or 2.
4. Any history of adverse events associated with cannabis intoxication or dependence.
5. A subject that has used one of the forbidden drugs, substances or foods as follows:

   * Any investigational product (THC or/and CBD ingestion or smoking) within one month preceding the study.
   * Any prescription or non-prescription medication (including herbal remedies, vitamins or dietary supplements) or vaccine within 14 days of the first day of study drug administration (Day 1) or within 5 half-lives before the first day of study drug administration, whichever is longer.

   Exceptions are locally acting medications (eg, topical creams), which are not allowed within 5 days of study drug administration, and the occasional use of acetaminophen (up to 3 g/day) and ibuprofen (up to 1200 mg/day).
   * Consumption of grapefruit, grapefruit juice, Seville oranges, pomelo containing products, within the 14 days prior to Day -1 and then throughout the entire study.
   * Consumption of excessive amounts of alcoholic beverages, defined as >3 drinks per day (beer, wine, or distilled spirits), or unwilling to comply with the restricted use of alcohol during the study (48 hours prior to admission and throughout the study), who have history of alcoholism.
6. Subject that has any condition that may possibly interfere with drug absorption, distribution, metabolism, or excretion (eg, previous surgery on the gastrointestinal tract [including removal of parts of stomach, bowel, liver, gall bladder, or pancreas] or stomach banding).
7. Exhausting physical exercise 48 hours prior to drug administration.
8. The subject does not agree to abstain from excessive caffeine and xanthine containing foods and beverages (ie, equivalent to >4 cups brewed coffee per day) from 48hr prior to Day -1 and throughout the entire study.
9. Those who had donated >0.5 L blood within 30 days of study.
10. Abnormal blood pressure and heart rate values according to the following criteria:

    * The subject has a supine pulse rate outside of the range of 40 to 100 bpm (following at least a 10-minute rest) measured at screening or Day -1.
    * The subject has a supine blood pressure outside of the range of 90 to 139 mm Hg systolic or 50 to 89 mm Hg diastolic (following at least a 10 minute rest) measured at screening or Day-1. Note: The blood pressure measurement may be repeated up to 3 times to meet eligibility requirements. In this case, the average of these 3 measurements must meet eligibility criteria.
11. A subject with a clinically significant history of drug allergies (including cannabis extracts, ethanol, or sesame oil), drug hypersensitivity or history of idiosyncratic reactions to any drug.
12. History of abuse of any drug/chemical.
13. Inability to relate to and/or cooperate with the investigators.
14. A subject with any other condition, which, in the opinion of the investigator, makes the subject inappropriate for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02-19 (Estimated); Study Completion 2025-02-19 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of CBD | 24 Hours
  Assesment of the pharmacokinetic profile of Cannabidiol in healthy volunteers. Plasma concentrations will be determined using HPLC-MS/MS validiated assay. The unit of measure will be provided as ng/ml.

SECONDARY OUTCOMES:
Exposure to the metabolites of the study drugs | 24 hours
  Assessment of the metabolic profile of the major cannabidiol metabolites: 7-hydroxy-CBD and CBD-glucoronide-11 in healthy volunteers. Plasma metabolites concentrations will be determined using HPLC-MS/MS validiated assay. The unit of measure will be provided as ng/ml.
Measurement of pharmacodynamic (PD) variables following CBD administration | 24 hours
  Cold pressor test - volunteers are requested to immerse their hands in ice cold water for up to two minutes. During the assesment the participants are requested to rate their pain scores from 0-100, at 15 second intervals for the duration of the two minute test time.
  In the event that the participant should remove their hands at any point during the assessment the VAS score is rated 100.
  This assesment is repeated muliple times for each participant throughout each study cycle.
Measurment of reaction time and coordination following CBD administration. | 24 hours
  Aim trainer test- A computerized eye hand coordination test to assess the response time and coherence following CBD administration. This test will be repeated multiple throughout each CBD administration cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Elyad Davidson, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel